CLINICAL TRIAL: NCT04127318
Title: Evaluating the Effects of Low-moderate Intensity Pedaling During Immunotherapy Administration on Immune Biomarkers and Quality of Life
Brief Title: Low-moderate Intensity Pedaling During Immunotherapy Administration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of resources
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19071102
Record Dates: First submitted 2019-09-26; First posted 2019-10-15 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Cancer of Skin; Cancer of Kidney; Cancer of Bladder; Exercise, Aerobic; Immunotherapy
Keywords: Sarcopenia; Quality of Life; Immunologic Markers
MeSH Terms: conditions — Skin Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms; Motor Activity; Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pedaling Group (Experimental): During their 30 minute immunotherapy infusions, participants will pedal using a stationary cycle ergometer. Participants will be allowed to determine their pedaling intensity and cadence, however, will be encouraged to reach the established goal intensity level. A research personnel will monitor the patient's heart rate, blood pressure, and RPE at baseline and every 10 minutes throughout the pedaling session. Participants will also have treatment response biomarkers gathered at baseline and before and within 10 minutes of completing their first and fourth immunotherapy infusions. Lastly, participants will complete both a physical activity questionnaire and a quality of life questionnaire at baseline and following their fourth treatment.
  Interventions: Behavioral: Pedaling Group

INTERVENTIONS:
Behavioral: Pedaling Group — Participants will pedal at low-moderate intensity using a stationary pedal ergometer concurrent to their immunotherapy infusion (30 minutes).

SUMMARY:
The purpose of this study is to determine the feasibility pedaling using an under-the desk bike during immunotherapy infusions. Also, the study hopes to evaluate how pedaling impacts quality of life and treatment response biomarkers. Lastly, the study will evaluate the relationships between treatment response and muscle mass which is evaluated with computerized tomography (CT) scans.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18
* Renal Cell Carcinoma, cutaneous malignancies (Melanoma, Merkel Cell Carcinoma or Squamous Cell CA) or bladder cancer.
* Planned intravenous immunotherapy treatment (Pembrolizumab, Nivolumab, or combinations as clinically indicated by standards of care).
* ECOG Performance Status of Grade 0-2
* No uncontrolled cardiac disease

Exclusion Criteria:

* ECOG Performance Status of Grade 3-5
* Severe cardiac history or comorbidities (i.e. heart failure, clinically significant aortic stenosis, history of cardiac arrest, have a cardiac defibrillator, uncontrolled angina, uncontrolled arrhythmias, major heart surgery, stroke, or pulmonary embolus).
* Chest pain or severe shortness of breath at rest or with physical activity.
* Orthopedic impediments to exercise (i.e. joint immobility or lower extremity lymphedema).
* Limitations to sustained exercise (i.e. bone metastases in the femur neck).
* Severe arthritis (i.e. osteoarthritis or rheumatoid arthritis).
* Patients will be excluded from study if their immunotherapy treatment requires the use of sedating antihistamines prior to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Pedaling Concurrent to Immunotherapy Infusions | 12 weeks
  The number of completed pedaling sessions as well as the ability of patients to meet goal pedaling intensities will be evaluated.

SECONDARY OUTCOMES:
Quality of life scores | 12 weeks
  Quality of life markers will be assessed using the Quality of Life Questionnaire - Core 30, at baseline and following their fourth immunotherapy treatment.
Treatment response biomarkers | 12 weeks
  Treatment response biomarkers (check point inhibitors, functional T and B cell subsets, pro and anti-inflammatory monocyte subsets, and soluble inflammatory mediators) will be drawn before and immediately following first and fourth immunotherapy treatments. All biomarkers are available as either part of the MILLIPLEX® MAP Human High-sensitivity T-cell Assay or the ProcartaPlex Human Immuno-Oncology Checkpoint Panel. All assays will be run according to the manufacturer's recommended protocols on a Luminex FlexMAP 3D system with concentrations calculated based on 7-point standard curves.
CT-derived sarcopenia rates | 12 weeks
  CT images will be gathered at the time of diagnosis and following completion of immunotherapy treatments. Patient's CT scans will be uploaded to a medical image analysis software (SliceOmatic), which allows for the evaluation of body composition, focusing on sarcopenia or muscle depletion.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Kuzel, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States